CLINICAL TRIAL: NCT00632671
Title: Constitution of a Population-based Cohort of Obese Subjects With Longitudinal Long-term Follow-up.
Brief Title: COLOMBES Project:Constitution of a Population-based Cohort of Obese Subjects With Longitudinal Long-term Follow-up
Acronym: COLOMBES
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P040807; AOM04013 (Other: french ministry)
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Obesity
Keywords: Obesity cohort
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, DNA, RNA, cell blood, for persons undergoing bariatric surgery (specific consentment): samples of liver and adipocytes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese persons cohorte: constitution of a prospective data collection (biological, clinical, paraclinical and questionnaires) in morbidly obese persons.

SUMMARY:
The objective of the project is the constitution of a population-based cohort of 500 persons with severe or morbid obesity (BMI over 35 kg/m2) with annual follow-up for 10 years. It aims to improve the physiopathological, epidemiological and prognostic knowledge of obesity and its consequences. Clinical data, biological material, exams and questionaires will be collected and stored, allowing the realisation of research works, initiated by research teams from our hospital or from other settings.

DETAILED DESCRIPTION:
The objective of this observational study is the follow-up of a cohort of 500 adult persons with morbid obesity (BMI>35 kg/m2).

Clinical and paraclinical data, and biological samples (plasma, serum, DNA, RNA, cell blood, for persons undergoing bariatric surgery (specific consent): samples of liver and adipocytes) will be collected and stored during the follow-up visits. These visits take place at inclusion, at 6 months, twelve months and every year for ten years. The collection of parental DNA will be proposed when feasable for genetic studies.

Persons will be recruited for four years, with an expected number of 350 persons included, in the clinical research unit of Louis MOURIER university hospital (AP-HP).

Each person included will participate in the study for ten years. When included, patients agree to come every year to follow-up visits. They are informed that data collected will be used only for research on obesity and its health consequences.

ELIGIBILITY:
Inclusion Criteria:

* BMI>35

Exclusion Criteria:

* previous bariatric surgery
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Morbidly obese subjects
Sampling Method: Non-Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2005-03; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Rate of follow-up at annual visit | annual

SECONDARY OUTCOMES:
Assessment of knee arthrosis (pain and radiological exam), at inclusion and after loss-weight (comparison after one and two years of follow-up of patients that did or did not undergo bariatric surgery). | one and two years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Simon Msika, MD, PhD, Principal Investigator — Louis Mourier University Hospital (AP-HP)
Locations (1):
- Louis Mourier hospital (AP-HP), Colombes, France